CLINICAL TRIAL: NCT06316518
Title: The Effect of Mindfulness-Based Web-Based Stress Reduction Program Applied to Primigravidas on Perceived Stress Level in Pregnancy, Birth Self-Efficacy and Prenatal Attachment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, YILMAZ, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AIBU-HF-YS-01
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Pregnancy Related
Keywords: Self Efficacy; Mindfulness; pregnancy; Stress,

STUDY DESIGN:
Intervention Model Description: Two groups with a supportive care control groups
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness group (Experimental): Primigravidas randomly assigned to the experimental group will be given web-based mindfulness-based stress reduction trainings after pre-tests are applied.
  Interventions: Other: mindfulness group
- control group (Active Comparator): After the pre-tests were applied to the control group, routine nursing care will be given and post-test measurements will be made after 8 weeks.
  Interventions: Other: mindfulness group

INTERVENTIONS:
Other: mindfulness group — In the study, primigravidas will receive 8-module (8-week-long) trainings, each lasting approximately 45 minutes, 3 days a week.

SUMMARY:
The aim of this study is to investigate the effect of a mindfulness-based web-based stress reduction program applied to primigravidas on perceived stress level in pregnancy, birth self-efficacy and prenatal attachment.

DETAILED DESCRIPTION:
Pregnancy is a process in which physical and hormonal changes occur in the female body. During this period, women experience mood swings due to changes in hormonal and social roles. These changes may predispose some women to mental health problems. Due to physiological and psychological changes during pregnancy, pregnant women may experience some problems such as nausea, vomiting, fatigue, anxiety, stress and depression . It is important to show pregnant women that these are normal experiences and to adopt an accepting attitude towards these experiences.

Perceived stress during pregnancy can cause many negative effects on maternal and fetal health. Among the causes of perceived stress are being diagnosed with a risky pregnancy, the presence of danger symptoms during pregnancy, the occurrence of adverse conditions during pregnancy and uncertainties about the pregnancy process.

Birth self-efficacy is defined as the level of assurance that a mother can give birth by using her abilities successfully. Birth self-efficacy is a motivating factor for the mother to cope with childbirth. High self-efficacy can reduce fear of childbirth and lead to better birth outcomes.

Prenatal attachment is defined as the expectant mother's attachment to the fetus through her behavior during pregnancy, establishing a close relationship and interacting with it. Prenatal attachment is an important component of the concept of fetal protection with the mother's attitudes of recognizing, being with and protecting her baby. The bond between mother and fetus has a great impact on the social and emotional development of the baby. A significant part of the attachment between mother and fetus begins during pregnancy and increases within a month after birth.

Supportive interventions, when necessary, to reduce perceived stress in pregnant women are critical for the protection of women's overall health. One of the non-pharmacological interventions is a mindfulness-based stress reduction program. Due to the success of standardized mindfulness-based interventions, mindfulness-based interventions have rapidly spread in western psychology research and practice. Abdolalipour et al. In a systematic review and meta-analysis of ten studies in 2023, Abdolalipour et al. reported that mindfulness practice reduced fear of childbirth.

ELIGIBILITY:
Inclusion Criteria:

* Graduated from at least primary school
* Having a computer or a cell phone,
* Having access to the Internet,
* Being between the ages of 18-35,
* Being 18-24 weeks pregnant,
* Having a single healthy fetus,
* Being primigravida,
* Not having a risky pregnancy (such as placenta previa, preeclampsia, not having any systemic disease),
* Not participating in any childbirth preparation class
* Not having a neurological or psychiatric disease.

Exclusion Criteria:

* Voluntary withdrawal from the study
* Failure to complete the 8-module training for any reason
* Interruption of internet access and inability to communicate
* Termination of pregnancy for any reason
* Non-participation in the trainings given in the experimental group

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Pregnancy Stress Assessment Scale (PSAS) | Two months
  The initial scale consisting of 40 items was revised as 36 items as a result of the validity and reliability study conducted in Taiwan. The scale consists of seven (7) sub-dimensions and is 5-point Likert type. Each item is evaluated as (absolutely no (0), mild (1), moderate (2), severe (3), very severe (4)). The lowest score that can be obtained from the scale is 0 and the highest score is 144.
Self-Efficacy Scale for Normal Childbirth | Two months
  There are 9 items in the scale. For each item in the scale, scores from 0 to 10 are given and scored as 0 points = no confidence at all and 10 points = very confident. The lowest score that can be obtained from the Self-Efficacy Scale for Normal Birth is 0, while the highest score that can be obtained is 90. As the scores obtained from the self-efficacy scale increase, the degree of self-efficacy also increases.
Prenatal Attachment Inventory (PAI) | Two months
  The inventory consists of 21 items and is four-point Likert type. The items of the inventory are scored between 1 and 4 points as 1-Never, 2-Sometimes, 3-Frequently, 4-Always. A minimum of 21 and a maximum of 84 points can be obtained from the inventory. An increase in the score obtained from the inventory indicates an increase in the level of attachment.

IPD SHARING:
Plan to Share IPD: Undecided